CLINICAL TRIAL: NCT06260423
Title: The Effect of Clinical Experience on the Quality of Obturation and Periapical Changes of Teeth Treated With Matched Cones in Combination With Bioceramic Sealer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Taha Badr, Assistant lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18/1/2024
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Obturation
Keywords: single cone; single matched cone
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experienced dentist using lateral compaction with bioceramic sealer group. (Experimental): The canals in this group obturation were obturated by an Experienced dentist using lateral compaction with bioceramic sealer.
  Interventions: Procedure: Experienced dentist using lateral compaction with bioceramic sealer.
- Unexperienced dentist using lateral compaction with bioceramic sealer group. (Experimental): The canals in this group obturation were obturated by an Unexperienced dentist using lateral compaction with bioceramic sealer.
  Interventions: Procedure: Unexperienced dentist using lateral compaction with bioceramic sealer.
- Experienced dentist using Single cone with bioceramic sealer group. (Experimental): The canals in this group obturation were obturated by an Experienced dentist using Single cone with bioceramic sealer.
  Interventions: Procedure: Experienced dentist using Single cone with bioceramic sealer.
- Unexperienced dentist using Single cone with bioceramic sealer group. (Experimental): The canals in this group obturation were obturated by an Unexperienced dentist using Single cone with bioceramic sealer.
  Interventions: Procedure: Unexperienced dentist using Single cone with bioceramic sealer.

INTERVENTIONS:
Procedure: Experienced dentist using lateral compaction with bioceramic sealer. — Root canal treatment using bioceramic sealers.
  Arms: Experienced dentist using lateral compaction with bioceramic sealer group.
Procedure: Unexperienced dentist using lateral compaction with bioceramic sealer. — Root canal treatment using bioceramic sealers.
  Arms: Unexperienced dentist using lateral compaction with bioceramic sealer group.
Procedure: Experienced dentist using Single cone with bioceramic sealer. — Root canal treatment using bioceramic sealers.
  Arms: Experienced dentist using Single cone with bioceramic sealer group.
Procedure: Unexperienced dentist using Single cone with bioceramic sealer. — Root canal treatment using bioceramic sealers.
  Arms: Unexperienced dentist using Single cone with bioceramic sealer group.

SUMMARY:
Evaluation of the impact of clinical experience on the quality of obturation and periapical changes of clinical cases using lateral compaction with bioceramic sealers and matched cone obturation with bioceramic sealers both clinically and radiographically.

DETAILED DESCRIPTION:
The idea of using single cone obturation is not novel historically, silver points were used in conjunction with various sealers. It has the advantages of being simple, is easy to learn, quick and does not require any complicated armamentarium or devices. Furthermore, unlike lateral or vertical compaction no force is used, therefore minimizing the risks of dentinal cracks. Recently single cone obturation in combination with bioceramic sealers has been advocated as an alternative obturation technique and is rapidly gaining popularity among dentists. Some studies have demonstrated that the amount of the overall porosity of the single cone fillings is comparable to other techniques.

ELIGIBILITY:
Inclusion Criteria:

patients with symptoms of irreversible pulpitis without apical periodontitis related to the maxillary first premolar ranging from 20 to 40 years old and with separate roots were selected from patients referred to the diagnosis clinic, Faculty of dental medicine Al-Azhar University, Cairo, Boys branch.

Exclusion Criteria:

1. Patients with any systemic disorders.
2. Pregnancy.
3. teeth with positive response to palpation test
4. Non vital teeth.
5. Teeth with positive response to percussion test.
6. Teeth with mobility of grade II or III.
7. teeth with probing depth more than 3 mm.
8. Teeth with abnormal morphology.
9. Teeth with root curvatures more than 20 degree (according to Schneider's method).
10. Teeth with internal or external root resorption.
11. Teeth with vertical root fracture.
12. Teeth with open apices.
13. Teeth with any root canal type other than type I.
14. Patients with (VDS) test with score 4 or less. 15- teeth with fused roots or single root.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain assessment | 24 hours
  The postoperative pain assessment was done using the modified verbal descriptor scale as follows:
  None (Score0), Mild(Score1), Moderate (Score2), and severe (Score3).
Postoperative pain assessment | 48 hours
  The postoperative pain assessment was done using the modified verbal descriptor scale as follows:
  None (Score0), Mild(Score1), Moderate (Score2), and severe (Score3).
Postoperative pain assessment | 72 hours
  The postoperative pain assessment was done using the modified verbal descriptor scale as follows:
  None (Score0), Mild(Score1), Moderate (Score2), and severe (Score3).
Postoperative pain assessment | 96 hours
  The postoperative pain assessment was done using the modified verbal descriptor scale as follows:
  None (Score0), Mild(Score1), Moderate (Score2), and severe (Score3).
Postoperative pain assessment | 120 hours
  The postoperative pain assessment was done using the modified verbal descriptor scale as follows:
  None (Score0), Mild(Score1), Moderate (Score2), and severe (Score3).

SECONDARY OUTCOMES:
The quality of obturation and the voids within the root canal filling | 24 hours
  the quality of obturation and the voids within the root canal filling were evaluated using Modified Coll and Sadrian criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar university, Cairo, Egypt